CLINICAL TRIAL: NCT00699816
Title: Randomized, Open-label, Multi-center and Phase 3 Clinical Trial to Compare the Efficacy and Safety of 'Green Cross CELL Immuncell-LC Group' and 'Non-treatment Group' in Patient Undergone Curative Resection(PEIT, RFA or Operation) for Hepatocellular Carcinoma in Korea
Brief Title: Efficacy and Safety of Immuncell-LC Group and Non-treatment Group in Hepatocelluar Carcinoma Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GC Cell Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIC-I01
Record Dates: First submitted 2008-06-17; First posted 2008-06-18 (Estimated); Results first posted 2015-09-24 (Estimated); Last update posted 2023-07-11 (Actual); Status verified 2015-08

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immunotherapy Group (Experimental): Adjuvant adoptive immune therapy using a CIK cell agent(Immuncell-LC) 16 times(4 treatments at a frequency of once per week, followed by 4 treatments every 2 weeks, then 4 treatments every 4 weeks, and finally 4 treatments every 8 weeks.
  Interventions: Biological: Immuncell-LC
- Control Group (No Intervention): Patients who had undergone curative treatment(surgical resection, radiofrequency ablation[RFA], or percutaneous ethanol injection[PEI]) for HCC of pretreatment clinical stage I or II according to the American Joint Committee on Cancer staging system(6th edition) based on radiologic imaging studies were eligible for this study with no adjuvant treatment

INTERVENTIONS:
Biological: Immuncell-LC — Activated T lymphocyte
  Arms: Immunotherapy Group

SUMMARY:
To prove that the efficacy and safety of 'Green Cross CELL* Immuncell-LC group' is superior to 'non-treatment group(Control group)' in patient undergone curative resection(PEIT, RFA or operation) for hepatocellular carcinoma in Korea

DETAILED DESCRIPTION:
Multicenter, randomized, open-labeled phase 3 clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Prior to the test, patient is fully explained about the purpose/ contents and characteristics of the testing medication, and the patient him(her)self, the guardian or the legal representative signed on written consent.
* The patient is more than 20 and less than 80 years old
* The patient is diagnosed as hepatocellular carcinoma by pathological/ radiological test and he (she) is in the stage of I or II. (refer to the attached file 10). Hepatocellular carcinoma should be shown by radiological test; on dynamic CT, dynamic MRI or on angiography.
* Child-Pugh Score should be less than 6 (refer to the attached file 7)
* No matter how the patient has been treated before, his (her) tumor should be totally removed by curative resection (PEIT, RFA or operation) in 12 weeks. (based on the agreement date for written consent) The tumor's removal should be perfectly confirmed by pathological or radiological test with the mentioned method in 3) at least 4 weeks later.
* ECOG Performance status (ECOG-PS) is less than 1 or equal to (refer to the exhibit 8)
* Patient's remaining life-time should be expected at least more than 3 months.
* Patient should meet below conditions by blood test, kidney and liver function test

  : Re-evaluation is possible during screening
* Leukocyte count is bigger than (3 multiply 109/L)
* Absolute Neutrophil Count (ANC) is bigger than or equal to 1,000/µL
* Hemoglobin is bigger than or equal to 8.5 g/dL
* Thrombocyte count is bigger than (5 multiply 1010/L)
* BUN and serum Creatinine is less than or equal to 1.5 multiply normal upper-limit
* No more disease abdominal extrahepatic transfer is confirmed by abdominal CT/ MRI

Exclusion Criteria:

* Hepatocellular carcinoma has been transferred by pathological/ radiological test (Stage III or Stage IV, refer to the exhibit 10)
* The carcinoma has been invaded to main portal vein or major branch hepatic vein
* Child-Pugh score is over 6
* Patient has serious problem with pulmonary function by sub- investigator's opinion
* Patient who has disease history of immune deficiency (which can be worse by immunotherapy) or auto-immune disease (ex. arthritis rheumatism, Burger's disease, multiple sclerosis and adolescent-occurred insulin dependent diabetes)
* Diagnosed as an immune deficiency patient
* Patient who has disease history of malignant tumor within 5 years before this clinical trial. (except for skin cancer, local prostate cancer or carcinoma in situ of the uterine cervix
* Patient who had anti-cancer medication before the clinical trial
* Patient who has serious disease in other organs after tumor resection.
* Patient has serious allergic-history by sub- investigator's opinion
* Patient has serious mental disease by sub- investigator's opinion
* Pregnant women, nursing mother or having intention of being pregnant during the clinical test
* Patient who participated in other clinical trial within 4 weeks before this clinical trial
* Patient who is incongruent to this clinical trial by sub- investigator's opinion.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2008-07; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jung Hwan Yoon, MD, Principal Investigator — Seoul National University Hospital
Locations (5):
- South Korea (5):
  - Korea University Ansan Hospital, Ansan-si, Gojan1-dong/Danwon-gu
  - Korea University Guro Hospital, Seoul, Guro 2-Dong, Guro-Gu
  - Samsung Medical Center, Seoul, Ilwon-dong/Gangnam-gu
  - Seoul Asan Medical center, Seoul, Pungnab2-dong/Songpa-gu
  - Seoul National University Hospital, Seoul, Yeongun-dong/Jongro-gu

REFERENCES:
- [Background] Takayama T, Sekine T, Makuuchi M, Yamasaki S, Kosuge T, Yamamoto J, Shimada K, Sakamoto M, Hirohashi S, Ohashi Y, Kakizoe T. Adoptive immunotherapy to lower postsurgical recurrence rates of hepatocellular carcinoma: a randomised trial. Lancet. 2000 Sep 2;356(9232):802-7. doi: 10.1016/S0140-6736(00)02654-4. PMID 11022927
- [Derived] Lee JH, Lee JH, Lim YS, Yeon JE, Song TJ, Yu SJ, Gwak GY, Kim KM, Kim YJ, Lee JW, Yoon JH. Adjuvant immunotherapy with autologous cytokine-induced killer cells for hepatocellular carcinoma. Gastroenterology. 2015 Jun;148(7):1383-91.e6. doi: 10.1053/j.gastro.2015.02.055. Epub 2015 Mar 4. PMID 25747273

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This phase 3 clinical study was a multicenter, randomized, open-labeled trial. The study was conducted at 5 university affiliated hospitals in Korea. All eligible participants were assigned randomly, in a 1:1 ratio, to receive adjuvant adoptive immune therapy using a CIK cell agent or no adjuvant treatment.
Groups:
- Immunotherapy Group: Patients who had undergone curative treatment(surgical resection, radiofrequency ablation[RFA], or percutaneous ethanol injection[PEI]) for HCC of pretreatment clinical stage I or II according to the American Joint Committee on Cancer staging system(6th edition) based on radiologic imaging studies were eligible for this study with adjuvant adoptive immune therapy using a CIK cell agent
Period: Overall Study
Arm/Group | Immunotherapy Group | Control Group
Started | 115 | 115
Completed | 114 | 112
Not Completed | 1 | 3
Not completed — Protocol Violation | 1 | 3

BASELINE CHARACTERISTICS:
Population: A total of 230 eligible participants were assigned randomly to either the immunotherapy group(n=115) or the control group(n=115). Among these randomized patients, 226(114 in the immunotherapy group and 112 in the control group) were included in the efficacy analysis. 4 patients were excluded due to violation of the inclusion and exclusion criteria.
Groups:
- Total: Total of all reporting groups
Arm/Group | Immunotherapy Group | Control Group | Total
Number analyzed (Participants) | 114 | 112 | 226
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 55.4 (8.2) | 56.4 (10.6) | 55.9 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 21 | 40
  Male | 95 | 91 | 186
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 114 | 112 | 226
Treatment modality [Number; unit: participants]
  Percutaneous ethanol injection | 13 | 4 | 17
  Radiofrequency ablation | 69 | 70 | 139
  Surgical resection | 32 | 38 | 70
HCC stage [Number; unit: participants] — HCC staging criteria is AJCC staging system(6th edition) developed by the American Joint Committee on Cancer for describing the extent of disease progression in cancer patients. It utilizes in part the TNM scoring system: Tumor size, Lymph Nodes affected, Metastases.
  The TNM Staging System is based on the extent of the tumor (T), the extent of spread to the lymph nodes (N), and the presence of metastasis (M). Once the T, N, and M are determined, they are combined, and an overall "Stage" of I, II, III, IV is assigned. Higher stage cancers are more advanced.
  participants
    Stage I | 98 | 94 | 192
    Stage II | 16 | 18 | 34
Number of HCC [Number; unit: participants] — Tumor assessments were performed using dynamic computed tomography or magnetic resonance imaging. All scans were reviewed by 2 independent radiologists at each site(hospital) with more than 5 years' experience, who were unaware of the group assignment. In cases of discordance, an additional third independent experienced radiologist reviewed images and consensus was achieved among the 3 radiologists.
  participants
    >3 or =3 | 2 | 2 | 4
    <3 | 112 | 110 | 222
Size of HCC [Median (Inter-Quartile Range); unit: centimeter] — Tumor assessments were performed using dynamic computed tomography or magnetic resonance imaging. All scans were reviewed by 2 independent radiologists at each site(hospital) with more than 5 years' experience, who were unaware of the group assignment. In cases of discordance, an additional third independent experienced radiologist reviewed images and consensus was achieved among the 3 radiologists.
  centimeter | 1.8 [1.4 to 2.3] | 2.3 [1.5 to 3.1] | 2.0 [1.4 to 2.7]
ECOG performance status [Number; unit: participants] — ECOG (Eastern Cooperative Oncology Group) performance status assesses the daily living abilities of the patient, on a scale ranging from 0(fully active) to 5(dead).
  participants
    0 | 81 | 81 | 162
    1 | 33 | 31 | 64
Cause of liver disease [Number; unit: participants]
  HBV infection only | 96 | 90 | 186
  HCV infection only | 9 | 10 | 19
  HBV and HCV | 2 | 2 | 4
  Co-infection (Others) | 7 | 10 | 17
  Co-infection (Cirrhosis) | 76 | 70 | 146
Alpha fetoprotein level [Median (Inter-Quartile Range); unit: ng/mL] | 5.2 [3.1 to 9.9] | 5.4 [3.0 to 13.0] | 5.3 [3 to 11.4]
PIVKA-II [Median (Inter-Quartile Range); unit: mAU/mL] | 19.0 [14.0 to 24.8] | 18.0 [14.0 to 24.0] | 18.5 [14 to 24.4]
Aspartate aminotransferase level [Median (Inter-Quartile Range); unit: IU/L] | 33.0 [27.0 to 43.5] | 34.0 [26.8 to 44.0] | 33.5 [26.9 to 43.8]
Alanine aminotransferase level [Median (Inter-Quartile Range); unit: IU/L] | 33.0 [25.0 to 45.8] | 33.0 [23.0 to 47.5] | 33.0 [24.0 to 46.7]
Alkaline phosphatase level [Median (Inter-Quartile Range); unit: IU/L] | 82.5 [70.0 to 101.5] | 82.0 [65.0 to 100.0] | 82.3 [67 to 100.3]
Albumin level [Median (Inter-Quartile Range); unit: g/dL] | 4.1 [3.9 to 4.3] | 4.1 [3.9 to 4.3] | 4.1 [3.9 to 4.3]
Total bilirubin level [Median (Inter-Quartile Range); unit: mg/dL] | 0.8 [0.6 to 1.0] | 0.8 [0.6 to 1.0] | 0.8 [0.6 to 1.0]
Prothrombin time [Median (Inter-Quartile Range); unit: seconds] | 13.7 [13.1 to 14.7] | 13.9 [13.2 to 14.4] | 13.8 [13.2 to 14.6]
Creatinine level [Median (Inter-Quartile Range); unit: mg/dL] | 0.9 [0.8 to 1.0] | 0.9 [0.7 to 1.0] | 0.9 [0.8 to 1.0]
Platelet [Median (Inter-Quartile Range); unit: x 10^3/mm^3] | 116.5 [92.3 to 158.0] | 141.0 [117.5 to 166.3] | 128.6 [100.0 to 157.2]

OUTCOME MEASURES:

1. Primary Outcome: Recurrence Free Survival(RFS)
Description: RFS was measured from the date of randomization to the first recurrence or to death from any cause.
Time Frame: Every 3months from the baseline for 24 months and then every 3-6 months until the data cut-off date, up to LSLV(Last Subject Last Visit)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Immunotherapy Group | Control Group
Number analyzed (Participants) | 114 | 112
months | 44.0 [42.46 to 44.54] | 30.0 [28.25 to 31.75]
Statistical Analysis 1: Comparison: Immunotherapy Group vs Control Group; Test type: Superiority or Other; p = 0.01, Log Rank; Hazard Ratio (HR) = 0.63, 95% CI 2-sided [0.43 to 0.94]

2. Secondary Outcome: Overall Survival(OS)
Description: Overall survival was measured from the date of randomization until death from any cause.
Time Frame: Every 3months from the baseline for 24 months, and then every 3-6 months until the data cut-off date, up to LSLV(Last Subject Last Visit)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Immunotherapy Group | Control Group
Number analyzed (Participants) | 114 | 112
months | NA [NA to NA] — At the time of the date cut-off date, 15 deaths had occurred in the efficacy population. Median OS was not reached. | NA [NA to NA] — At the time of the date cut-off date, 15 deaths had occurred in the efficacy population. Median OS was not reached.
Statistical Analysis 1: Comparison: Immunotherapy Group vs Control Group; Test type: Superiority or Other; p = 0.008, Log Rank; Hazard Ratio (HR) = 0.21, 95% CI 2-sided [0.06 to 0.75]

3. Secondary Outcome: Cancer-specific Survivals
Description: Cancer-specific survival was measured from the date of randomization until death resulting from HCC.
Time Frame: Every 3 months from baseline for 24 months, and then every 3-6 months until the data cut-off date, up to LSLV(Last Subject Last Visit)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Immunotherapy Group | Control Group
Number analyzed (Participants) | 114 | 112
months | NA [NA to NA] — At the time of the date cut-off date, 15 deaths had occurred in the efficacy population. Median Cancer-specific survival was not reached. | NA [NA to NA] — At the time of the date cut-off date, 15 deaths had occurred in the efficacy population. Median Cancer-specific survival was not reached.
Statistical Analysis 1: Comparison: Immunotherapy Group vs Control Group; Test type: Superiority or Other; p = 0.02, Log Rank; Hazard Ratio (HR) = 0.19, 95% CI 2-sided [0.04 to 0.87]

4. Primary Outcome: Recurrence Free Survival(RFS) Rate
Description: RFS rate was measured from the date of randomization to the first recurrence or to death from any cause.
Time Frame: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Immunotherapy Group | Control Group
Number analyzed (Participants) | 114 | 112
percentage of participants
  RFS rate 12 months | 79.9 | 65.1
  RFS rate 24 months | 72.5 | 53.8
  RFS rate 36 months | 60.9 | 44.3
  RFS rate 48 months | 49.6 | 39.6

5. Secondary Outcome: Overall Survival(OS) Rate
Description: Overall survival rate was measured from the date of randomization until death from any cause.
Time Frame: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Immunotherapy Group | Control Group
Number analyzed (Participants) | 114 | 112
percentage of participants
  OS rate 12 months | 100.0 | 98.0
  OS rate 24 months | 100.0 | 91.8
  OS rate 36 months | 97.5 | 88.1
  OS rate 48 months | 95.9 | 84.8

6. Secondary Outcome: Cancer-specific Survival Rate
Description: Cancer-specific survival rate was measured from the date of randomization until death resulting from HCC.
Time Frame: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Immunotherapy Group | Control Group
Number analyzed (Participants) | 114 | 112
percentage of participants
  Cancer-specific survival rate 12 months | 100.0 | 98.0
  Cancer-specific survival rate 24 months | 100.0 | 94.9
  Cancer-specific survival rate 36 months | 98.8 | 91.0
  Cancer-specific survival rate 48 months | 97.2 | 87.5

ADVERSE EVENTS:
Time Frame: Adverse events were assessed from the time the patient provided written informed consent until the end of the study or drop-out, and until at least 30 days after the last dose of immunotherapy.
Arm/Group | Immunotherapy Group | Control Group
Serious Adverse Events (participants affected / at risk) | 9/115 | 4/115
Other Adverse Events (participants affected / at risk) | 71/115 | 47/115
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immunotherapy Group (N=115) | Control Group (N=115)
Sudden hearing loss (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Meniscus lesion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
High frequency ablation (Surgical and medical procedures) | 1 (1) | 0 (0)
Hepatic vein stenosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immunotherapy Group (N=115) | Control Group (N=115)
Upper respiratory tract infection (Infections and infestations) | 6 (6) | 4 (5)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Body tinea (Infections and infestations) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (5) | 4 (4)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 5 (5)
Sudden hearing loss (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 11 (24) | 0 (0)
Pyrexia (General disorders) | 12 (22) | 0 (0)
Dizziness (Nervous system disorders) | 5 (5) | 3 (3)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 3 (4)
Herpes zoster (Infections and infestations) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (6) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 6 (6) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 11 (12) | 3 (3)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Epigastric discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 1 (1)
Chest discomfort (General disorders) | 3 (3) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 2 (2)
Gastritis erosive (Gastrointestinal disorders) | 1 (1) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (1) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 2 (4) | 2 (3)
Gastritis (Gastrointestinal disorders) | 0 (0) | 3 (3)
Gastric polyps (Gastrointestinal disorders) | 0 (0) | 3 (3)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (4) | 2 (2)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 3 (3)
Headache (Nervous system disorders) | 3 (4) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 3 (3)
Weight increased (Investigations) | 2 (3) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No